CLINICAL TRIAL: NCT06130072
Title: Hysteroscopic Tubal Occlusion Using Iso-amyl- 2-cyanoacrylate With or Without Ethiodized Oil (Lipidol) in Patients With Hydrosalpinx Prior to IVF
Brief Title: Hysteroscopic Tubal Occlusion Using Amacrylate With or Without Lipidol in Patients With Hydrosalpinx Prior to IVF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed I Amer, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ASU124
Record Dates: First submitted 2023-10-28; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Effectiveness of Isoamyl-2-cyanoacrylate With and Without Ethiodized Oil in Occluding Hydrosalpinx Prior to IVF
MeSH Terms: interventions — Ethiodized Oil

STUDY DESIGN:
Intervention Model Description: Hysteroscopic tubal occlusion using iso-amyl- 2-cyanoacrylate with or without Ethiodized oil (Lipidol) in patients with hydrosalpinx prior to IVF
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopic tubal occlusion using iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil (Active Comparator): Group 2 including 20 patients with hydrosalpinx refaired for hysteroscopic tubal occlusion prior to IVF using iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil.
  Interventions: Drug: iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil
- Hysteroscopic tubal occlusion using only iso-amyl- 2-cyanoacrylate (Active Comparator): Group 1 including 25 patients with hydrosalpinx refaired for hysteroscopic tubal occlusion prior to IVF using iso-amyl- 2-cyanoacrylate .
  Interventions: Drug: iso-amyl- 2-cyanoacrylate.

INTERVENTIONS:
Drug: iso-amyl- 2-cyanoacrylate. — Hysteroscopic tubal occlusion using iso-amyl- 2-cyanoacrylate in patients with hydrosalpinx prior to IVF
  Arms: Hysteroscopic tubal occlusion using only iso-amyl- 2-cyanoacrylate
Drug: iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil — iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil (Lipidol)
  Arms: Hysteroscopic tubal occlusion using iso-amyl- 2-cyanoacrylate mixed with Ethiodized oil

SUMMARY:
Hysteroscopic tubal occlusion using iso-amyl- 2-cyanoacrylate with or without Ethiodized oil (Lipidol) in patients with hydrosalpinx prior to IVF

DETAILED DESCRIPTION:
hysteroscopic injection of iso-amyl- 2-cyanoacrylate with or without Ethiodized oil (Lipidol) in patients with hydrosalpinx requiring IVF. after one months and two months of the primary injection hysterosalpingography will be done to test for tubal occlusion.

ELIGIBILITY:
Inclusion Criteria: • Infertile women due to tubal factor with hydrosalpinx (unilateral or bilateral) prepared for IVF

Exclusion Criteria:

* • Any patient with acute pelvic inflammatory disease, endometritis, lower genital tract infection.

  * The presence of intrauterine synechiae that might hinder the proper hysteroscopic examination and tubal cannulation diagnosed by diagnostic hysteroscopy.
  * The presence of uterine anomalies that might hinder the proper hysteroscopic examination and tubal cannulation diagnosed by diagnostic hysteroscopy.
  * Undiagnosed genital bleeding.

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Fallopian tube occlusion | one to three months
  hysteosaplingographic diagnosis of tubal occlusion